CLINICAL TRIAL: NCT04414488
Title: The Impact of Regional Anaesthesia on Hormone Levels in Thoracic Surgery.
Status: Completed | Type: Observational
Sponsor: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Piotr Palaczyński, Principal Investigator, Medical University of Silesia
Other Study IDs: HL-01
Record Dates: First submitted 2020-05-30; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Hormones; Anesthesia, Conduction; Thoracic Surgical Procedure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient controlled analgesia: General anaesthesia was induced with midazolam 0.1 mg*kg-1, propofol 2 mg*kg-1, cisatracurium 0.15 mg*kg-1 and fentanyl 1.5 µg*kg-1. Anaesthesia was maintained with one minimal alveolar concentration sevoflurane. Fractional doses of fentanyl 1-3 µg*kg-1 were administered if heart rate or mean blood pressure rose more than 20% above the base-line value obtained just before surgery commenced. After surgery, if a patient complained of pain then she/he was given i.v. oxycodone by an anaesthetist before commencing the patient controlled analgesia (PCA). The PCA solution was oxycodone (1mg*ml-1) and the PCA was programmed to allow a self-administered bolus dose of 1mg oxycodone with a lockout time of 5 min. During the night, basal rate oxycodone was 2-4 mg per hour. Additionally, patients were given 1g intravenous paracetamol every 6h and 100mg of intravenous ketoprofen every 12h, if required.
- Thoracic paravertebral block and patient controlled analgesia: Before induction of general anesthesia thoracic paravertebral block was performed. General anaesthesia was induced with midazolam 0.1 mg*kg-1, propofol 2 mg*kg-1, cisatracurium 0.15 mg*kg-1 and fentanyl 1.5 µg*kg-1. Anaesthesia was maintained with one minimal alveolar concentration sevoflurane. Fractional doses of fentanyl 1-3 µg*kg-1 were administered if heart rate or mean blood pressure rose more than 20% above the base-line value obtained just before surgery commenced. After surgery, if a patient complained of pain then she/he was given i.v. oxycodone by an anaesthetist before commencing the patient controlled analgesia (PCA). The PCA solution was oxycodone (1mg*ml-1) and the PCA was programmed to allow a self-administered bolus dose of 1mg oxycodone with a lockout time of 5 min. During the night, basal rate oxycodone was 2-4 mg per hour. Additionally, patients were given 1g intravenous paracetamol every 6h and 100mg of intravenous ketoprofen every 12h, if required.
  Interventions: Procedure: Thoracic paravertebral block (ThPVB)

INTERVENTIONS:
Procedure: Thoracic paravertebral block (ThPVB) — Before the induction of general anaesthesia a single-shot ThPVB was performed at the Th3 to Th4 level, approximately, 2.5 to 3 cm lateral to tip of a spinous process. A preblock ultrasound examination was undertaken to assess the depth of the transverse process and the pleura. An insulated 10 cm long needle was used and this was connected to a peripheral nerve stimulator with a set current of 2.5 milliampere(mA). The current was gradually reduced as the needle was inserted until the appearance of visible intercostal muscles activity with a current of 0.3 to 0.5mA (paravertebral space identification). Plain bupivacaine (0.3 ml*kg-1) was then injected after a negative aspiration test for air or blood. The efficacy of the blockade to cold was checked after 20 min with a plastic ampoule of saline kept in the freezer. Testing was symmetrical on both sides of thorax. A difference in sensation to cold between the blocked and unblocked sides was taken to indicate an effective block.
  Groups: Thoracic paravertebral block and patient controlled analgesia

SUMMARY:
Basic aspects of thoracic anaesthesia are general anesthesia often combined with regional anesthesia, intubation with double lumen tube and separation of lung ventilation. Proper assessment of pain and adequate analgesia in intraoperative and postoperative period is a challenging issue for medical practitioners. Intraoperative trauma may lead to many metabolic implications and disturbance of haemostasis, what can be reflected in change of blood and saliva hormone and other substance levels. The aim of this study is to assess the impact of regional anesthesia on hormone levels in patients requiring videothoracoscopic procedures.

DETAILED DESCRIPTION:
Basic aspects of thoracic anaesthesia are general anesthesia often combined with regional anesthesia, intubation with double lumen tube and separation of lung ventilation. Proper assessment of pain and adequate analgesia in intraoperative and postoperative period is a challenging issue for medical practitioners. Intraoperative trauma may lead to many metabolic implications and disturbance of haemostasis, what can be reflected in change of blood and saliva hormone and other substance levels, such as alpha-amylase, cortisol, testosterone, secretory IgA, β-endorphin, nerve growth factor, calcitonin gene-related protein and P substance. The aim of this study is to assess the impact of regional anesthesia on hormone levels in postoperative period. Saliva was collected from participants in order to perform laboratory tests, using a special disposable Salivette tube (Sarstedt AG & Co, Germany). Saliva was collected by placing a sterile tampon under the tongue or chewing for 30-45 seconds. The soaked saliva pad was then placed in a suspended insert with a perforated bottom. The insert with a tampon was placed in a centrifuge tube and closed with a stopper. Next the tube was centrifuged (1000 x g for 10 min.) to obtain a ready to test saliva supernatant. Approximately 0,7 ml of the supernatant from every sample collected was used for further testing. Samples were frozen after centrifugation at - 85°C until performing laboratory tests. Blood was collected for laboratory tests from the ulnar vein. Blood for testing was collected using disposable equipment in a volume of 5ml into a tube containing ethylenediaminetetraacetic acid (EDTA) and aprotinin. Next the tube was centrifuged (1000 x g for 5 min.). After centrifugation and separation of morphotic elements, the obtained plasma was divided into two tubes and frozen at - 85°C until performing laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

-qualification to elective videothoracoscopic procedures and general anaesthesia

Exclusion Criteria:

* lack of consent to participation in the study,
* significant coagulopathy,
* contraindication to the thoracic paravertebral block or drugs used in protocol,
* history of chronic pain,
* chest wall neoplastic invasion,
* previous thoracic spine surgery,
* mental state preventing from effective use of PCA device,
* renal failure (GFR <60 ml/min/1,73 m2).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population consisted of consecutive patients scheduled for elective videothoracoscopic procedures.
Sampling Method: Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Alpha-amylase activity. [U/ml] | 24 hours
  α-amylase activity assay was performed by a static method with AMYLAZA kit (Aqua-Med Łodz, Poland). The samples were diluted 100 times using 0,9% chloride solution. 2-chloro-4-nitrofenylo-maltotrioside is a substrate in this method. The reaction was performed in pH 6,0 MES buffer at 37 ° C rendering a colored reaction product. The product was then analyzed via spectrophotometry at 405 nm. Results are presented in salivary α-amylase activity units (U/ml). Measurement imprecision of the method was 4.1%. Material was collected after enrollment to the study (T0), six hours after the surgery (T1) and 24 hours after the surgery (T2).
Cortisol concentration. [ng/ml] | 24 hours
  The commercial ELISA (Diapra, Italy) was used to determine the concentration of cortisol. The analytical procedure was in accordance with the manufacturer's instructions in the technical manuals supplied with the kits. Absorbance readings were taken using a µQuant reader (Biotek, USA), while results were processed using KCJunior (Biotek, USA). The sensitivity of the method was 0,12 ng/ml for cortisol. The method's imprecision was 6.2%. Material was collected after enrollment to the study (T0), six hours after the surgery (T1) and 24 hours after the surgery (T2).
Testosterone concentration. [pg/ml] | 24 hours
  The commercial ELISA (Diapra, Italy) was used to determine the concentration of testosterone. The analytical procedure was in accordance with the manufacturer's instructions in the technical manuals supplied with the kits. Absorbance readings were taken using a µQuant reader (Biotek, USA), while results were processed using KCJunior (Biotek, USA). The sensitivity of the method was 3,28 pg/ml for testosterone. The method's imprecision was 7.9%. Material was collected after enrollment to the study (T0), six hours after the surgery (T1) and 24 hours after the surgery (T2).
Secretory Immunoglobulin A concentration. (sIgA) | 24 hours
  The commercial ELISA (Immunodiagnostic AG, Niemcy.) were used to determine the concentration of sIgA. The analytical procedure was in accordance with the manufacturer's instructions in the technical manuals supplied with the kits. Absorbance readings were taken using a µQuant reader (Biotek, USA), while results were processed using KCJunior (Biotek, USA). Material was collected after enrollment to the study (T0), six hours after the surgery (T1) and 24 hours after the surgery (T2).
β-endorphin concentration. | 24 hours
  Determination of β-endorphin concentration was preceded by extraction on C18 Sep-Pak columns containing 50mg C18, using trifluoroacetic acid (TFA) and elution buffer (i.e. 60% acetonitrile, 1% TFA and 39% distilled water). The extracts obtained were lyophilized. To determine the concentration of β-endorphins in the tested samples, lyophilisates were dissolved in an appropriate amount of buffer, and then commercial ELISA tests from Elabscience, USA were used. The analytical procedure was in accordance with the manufacturer's instructions in the technical manuals supplied with the kits. Absorbance readings were taken using a µQuant reader (Biotek, USA), while results were processed using KCJunior (Biotek, USA). Material was collected after enrollment to the study (T0), six hours after the surgery (T1) and 24 hours after the surgery (T2).
P substance concentration. [pg/ml] | 24 hours
  The commercial ELISA test was used to determine the concentration of P substance. The analytical procedure was in accordance with the manufacturer's instructions in the technical manuals supplied with the kits. Material was collected after enrollment to the study (T0), six hours after the surgery (T1) and 24 hours after the surgery (T2).
Nerve Growth Factor concentration. [ng/ml] | 24 hours
  The commercial ELISA test was used to determine the concentration of the Nerve Growth Factor. The analytical procedure was in accordance with the manufacturer's instructions in the technical manuals supplied with the kits. Material was collected after enrollment to the study (T0), six hours after the surgery (T1) and 24 hours after the surgery (T2).
Calcitonin Gene-related Peptide concentration. [pg/ml] | 24 hours
  The commercial ELISA test was used to determine the concentration of the Calcitonin Gene-related Peptide. The analytical procedure was in accordance with the manufacturer's instructions in the technical manuals supplied with the kits. Material was collected after enrollment to the study (T0), six hours after the surgery (T1) and 24 hours after the surgery (T2).

SECONDARY OUTCOMES:
Pain intensity (NRS) | 24 hours
  Pain intensity at rest was recorded with Numerical Rating Scale (NRS) at 0, 6, 12, 18 and 24 postoperative hours. Patient determined intensity of symptoms on a 10 grade scale, where 0 corresponded to no pain and 10 corresponded to the strongest possible pain.
Arterial blood pressure [mmHg] | 24 hours
  Non-invasive arterial blood pressure was recorded at 0, 6, 12, 18 and 24 postoperative hours.
Heart rate [bmp] | 24 hours
  Heart rate was recorded in continuous manner up to 24 postoperative hours.
Arterial blood saturation measured by pulse oximetry [%] | 24 hours
  Arterial blood saturation was recorded in continuous manner up to 24 postoperative hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Samodzielny Publiczny Szpital Kliniczny nr 1, Zabrze, Silesian Voivodeship, Poland